CLINICAL TRIAL: NCT03985553
Title: Development of a Self- Management Program for Parents With Spinal Cord Injury and Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Paralyzed Veterans of America (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201501151
Record Dates: First submitted 2019-05-30; First posted 2019-06-13 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Spinal Cord Injuries
Keywords: Parenting; Spinal Cord Injuries; Self-Management; Occupational Therapy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Parents/grandparents/potential parents with SCI/D had the opportunity to attend and participate in a 4 week self-management program once a week related to parenting with a disability. The self-management sessions lasted approximately 2 hours once a week and were led by an occupational therapist. There was no control group or alternate intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parenting Self-Management Program (Other): Participants were provided a Parenting Self -Management Program booklet with the twenty-four fact sheets at the beginning of the four-week program on topics such as adaptive babycare techniques, advocacy in the courts, emergency planning, safety in the community, talking to children about disability, managing pain/fatigue, connecting to other parents with SCI/D, and wheelchair adjustment/management during and after pregnancy. Sessions included topic introduction, participant interaction, goal setting, resource utilization, and program evaluation. Participants were allowed to choose which resources they wanted and what tips to incorporate into their parenting roles. Participants were asked to develop a weekly goal to encourage achievement, allowing individuals to identify what they wanted or decided to do that could be related to parenting directly or indirectly, such as health and wellness goals that gave them more energy or strength to complete parenting tasks.
  Interventions: Behavioral: Parenting Self-Management Program

INTERVENTIONS:
Behavioral: Parenting Self-Management Program

SUMMARY:
The purpose of this project was to develop and pilot test a self-management program targeted toward individuals with Spinal Cord Injury/Disease (SCI/D) who are current parents or who are considering becoming parents. This Parenting Self-Management Program (PSMP) will allow parents to identify their goals for successful family participation and provide a structure for professionals to use when working with parents with SCI/D to best meet their needs. A draft PSMP was assembled by members of the research team. This draft was reviewed by experienced parents with SCI/D and professionals who work with individuals who have SCI/D through key informant interviews or focus groups. The feedback was used to modify the draft program and the PSMP was pilot tested with a group of 10 individuals with SCI/D who are new parents, newly injured or who want to improve their participation in parenting activities.

DETAILED DESCRIPTION:
The project used a self-management approach grounded in self-efficacy theory to increase parenting self-efficacy among persons with spinal cord injury/disease (SCI/D). Program content focused on skill building through opportunities to master techniques and strategies; role modeling, problem solving, decision making, goal setting, and provision of reliable information. The use of a self-management program may also place parents with SCI/D at ease in sharing needs, as it is not an expert model by which a professional is passing judgment on their ability to care for their children. Many parents with disabilities are hesitant to seek professional services for fear of negative consequences such as losing custody of their children. Developing a program that is conducted as a partnership whereby parents direct much of the pace and content may be considered less threatening and more beneficial to those who have experienced distrust of the healthcare system.

There are no other self-management programs that specifically address the needs of parents with SCI/D. The project created a self-management program that was piloted in the St. Louis region and can be replicated across the country among other communities. While the national coordination center for families with disabilities, Through the Looking Glass, provides resource materials to parents across the country, they do not provide a structure for individual problem solving and to meet the needs of parents SCI/D on an individualized level. Providing a format for parents with SCI/D to successfully fulfill their parenting roles has a highly significant social implication; parents will be equipped to meet potential challenges and enjoy participation in their families. Limiting discrimination in the courts, seeking school accessibility, or simply decreasing pain while holding an infant are all worthy goals that could be achieved through a self-management parenting program.

Project Aims

1. To develop a four-week self-management program for parents with SCI/D to meet their needs in the parenting role and the needs of their families
2. To aid parents with SCI/D in building the skills and resources needed to continue or begin parenting in a successful manner
3. To disseminate the PSMP content to other regions, disability organizations, Paralyzed Veterans of America (PVA) chapters, healthcare organizations, and parenting groups to be replicated
4. To build a sustainable format for meeting the needs of parents with SCI/D that can be replicated and continued across the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older, parent/guardian/grandparent with diagnosis of SCI/D, community dwelling, able to read at or above sixth grade level and either newly injured (sustained SCI in last year) or self-identified as being less experienced in their parenting role.

Exclusion Criteria:

* Individuals were excluded if they were under age 18, did not have SCI/D, were not a parent/guardian/grandparent or lived in an institution.

A convenience sampling method was used to recruit participants through distribution of flyers at rehabilitation facilities, independent living centers and word of mouth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

PRIMARY OUTCOMES:
Change in participation using the Participation Survey- Mobility (PARTS-M) | Prior to first session of the PSMP group and 4 weeks after the initial session of the PSMP group.
  The PARTS/M is a reliable and valid self-report survey that assesses the participation of people with mobility limitations in various life activities and the impact of common environmental factors on participation (Gray, Hollingsworth, Stark, & Morgan, 2006). For the purposes of the PSMP, a modified version of the Parenting section of the PARTS/M was used. Participants were asked how often they participate in parenting activities, their evaluation of their participation (importance, choice, satisfaction, and control), the number and value of supports they may use, and the influence of pain and fatigue on their participation in parenting activities.
Change in self-efficacy using the General Self-Efficacy Scale (GSE) | Prior to first session of the PSMP group and 4 weeks after the initial session of the PSMP group.
  The GSE was used to determine any influence of the program on participants' self-efficacy. Total score ranges from 10-40 with higher values indicating better outcome.

SECONDARY OUTCOMES:
Demographic items | Prior to first session of the PSMP group and 4 weeks after the initial session of the PSMP group as needed.
  Age, gender, race, marital status, education level, living situation, income, benefits received, diagnosis associated with SCI/D, time with disability, additional impairments, secondary conditions (pain & fatigue), health status, mobility device use, personal assistance use
Parenting tasks | Prior to first session of the PSMP group
  Asked about number of children, ages, ages when acquired disability and open ended questions about most important and most difficulty task, use of strategies and assistance received when children were at various stages.
Skills and Knowledge | Prior to first session of the PSMP group and 4 weeks after the initial session of the PSMP group.
  Participants were asked to rate their knowledge of topics that were going to be included in the PSMP on a 0-10 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Dashner, OTD, Principal Investigator — Washington University Program in Occupational Therapy
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Results may be shared in the future following publication acceptance in peer reviewed journal. Individual data requests from researchers will be considered as needed at that time.

REFERENCES:
- [Background] Gray DB, Hollingsworth HH, Stark SL, Morgan KA. Participation survey/mobility: psychometric properties of a measure of participation for people with mobility impairments and limitations. Arch Phys Med Rehabil. 2006 Feb;87(2):189-97. doi: 10.1016/j.apmr.2005.09.014. PMID 16442971
- [Background] Bodenheimer T, Lorig K, Holman H, Grumbach K. Patient self-management of chronic disease in primary care. JAMA. 2002 Nov 20;288(19):2469-75. doi: 10.1001/jama.288.19.2469. PMID 12435261
- [Background] Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med. 2003 Aug;26(1):1-7. doi: 10.1207/S15324796ABM2601_01. PMID 12867348
- [Background] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Background] Nolte S, Elsworth GR, Sinclair AJ, Osborne RH. The extent and breadth of benefits from participating in chronic disease self-management courses: a national patient-reported outcomes survey. Patient Educ Couns. 2007 Mar;65(3):351-60. doi: 10.1016/j.pec.2006.08.016. Epub 2006 Oct 5. PMID 17027221
- [Background] O'Toole L, Connolly D, Smith S. Impact of an occupation-based self-management programme on chronic disease management. Aust Occup Ther J. 2013 Feb;60(1):30-8. doi: 10.1111/1440-1630.12008. Epub 2012 Nov 19. PMID 23414187
- [Background] Signore C, Spong CY, Krotoski D, Shinowara NL, Blackwell SC. Pregnancy in women with physical disabilities. Obstet Gynecol. 2011 Apr;117(4):935-947. doi: 10.1097/AOG.0b013e3182118d59. PMID 21422868
- [Background] Luszczynska A, Scholz U, Schwarzer R. The general self-efficacy scale: multicultural validation studies. J Psychol. 2005 Sep;139(5):439-57. doi: 10.3200/JRLP.139.5.439-457. PMID 16285214
- [Background] Barlow J, Wright C, Sheasby J, Turner A, Hainsworth J. Self-management approaches for people with chronic conditions: a review. Patient Educ Couns. 2002 Oct-Nov;48(2):177-87. doi: 10.1016/s0738-3991(02)00032-0. PMID 12401421